CLINICAL TRIAL: NCT01982409
Title: A Study of Immune Persistence After Inoculated With One-dose Freeze-dried Live Attenuated Varicella Vaccine in Children Aged 1-6 Years
Brief Title: Immune Persistence After Inoculated With One-dose Freeze-Dried Live Attenuated Varicella Vaccine in Children Vaccine in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Changchun Changsheng Life Science and Technology Co., Ltd. (Industry)
Collaborators: Guangdong Provincial Institute of Biological Products And Materia Medica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCT02038508
Record Dates: First submitted 2013-10-24; First posted 2013-11-13 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Chickenpox
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Live Attenuated Varicella Vaccine (Experimental): use the arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: Live Attenuated Varicella Vaccine

INTERVENTIONS:
Biological: Live Attenuated Varicella Vaccine

SUMMARY:
The purpose of this study is to observe the persistence of protection, duration of protection, safety and breakthrough infection rates afforded by live attenuated varicella vaccine in children over a 5-year period.

ELIGIBILITY:
Inclusion Criteria:

* Participant are healthy children aged 1-6 years, who has inquired for medical history and physical examination, and met the requirement of the vaccine trial
* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures
* Body temperature ≤37℃

Exclusion Criteria:

* Participant with previous history of chickenpox or zoster
* Receipt of varicella vaccine
* Reported the family history of allergies, convulsions, epilepsy and mental illness
* Known allergy to any constituent of the vaccine
* Known serve illness, in a fever, acute infection and chronic disease activity
* Receipt of steroid
* Reported the history of thrombocytopenia or other coagulation disorders, which may cause
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Known congenital malformation, developmental disorders and severe chronic disease (e.g. Down's syndrome, diabetes, sickle cell anemia and neurologic disorders)
* Known dermatopathy with allergy, herpes, fester, and fungal infection
* Receipt of whole blood, blood plasma or immunoglobulin in the 3 months preceding the trial vaccination
* Reported the history of acute illness had need systemic antibiotics or anti-viral treatment of infections in the 7 days preceding the trial vaccination
* Participant with fever(temperature≥ 38℃) in the days
* Any condition, which, in the opinion of the investigator, would pose a health risk to the subject

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2013-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Immune protective effect and persistence after inoculated with live attenuated varicella vaccine | Before vaccination, six weeks and every year in 5 years study period after inoculation of the live varicella vaccine
  Clinical subjects are drawn 3ml's vein blood，respectively before vaccination, six weeks and every year in 5 years study period after inoculation of the live varicella vaccine. FAMA methods are used to test antibody rate of pox virus.

SECONDARY OUTCOMES:
Breakthrough rate, duration and severity of varicella in vaccinated children | 5 years period
Occurrence of adverse events | Up to 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Maoming Center for Disease Control and Prevention, Maoming, Guangdong, China